CLINICAL TRIAL: NCT03921138
Title: Opportunistic Salpingectomy at the Time of Benign Laparoscopic Hysterectomy : Assessment of Possible Complications and Histopathological Tumor Protein 53 (p53)-Signatures
Brief Title: Opportunistic Salpingectomy at the Time of Benign Laparoscopic Hysterectomy
Acronym: SLH
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: SLH
Record Dates: First submitted 2019-04-16; First posted 2019-04-19 (Actual); Last update posted 2019-04-19 (Actual); Status verified 2019-04

CONDITIONS: Benign Laparoscopic Hysterectomy; Systematic Salpingectomy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Benign laparoscopic hysterectomy: Patients who underwent benign laparoscopic hysterectomy with systematic salpingectomy
  Interventions: Other: Histopathologic tube anomalies

INTERVENTIONS:
Other: Histopathologic tube anomalies — Assessment of prevalence of histopathologic tube anomalies (Serous Tubal Intraepithelial Carcinoma (STIC) or tumor protein 53 (p53) lesion)

SUMMARY:
In this prospective study, patients who underwent benign laparoscopic hysterectomy with systematic salpingectomy were included. The aim of this study is to assess the prevalence of tubal histopathological abnormalities such as Serous Tubal Intraepithelial Carcinoma (STIC) and tumor protein 53 (p53) signatures) as well as the prevalence of perioperative and postoperative complications related to opportunistic laparoscopic salpingectomy in a low risk population. The hypothesis is that prophylactic salpingectomy during benign laparoscopic hysterectomy is both feasible and innocuous. Peri- and postoperative complications, duration of salpingectomy and post-salpingectomy blood loss, histopathological and immunohistochemical analysis with anti-p53 antibody were evaluated.

ELIGIBILITY:
Inclusion Criteria:

* patients who underwent benign laparoscopic hysterectomy with systematic salpingectomy

Exclusion Criteria:

* Hysterectomy in a context of gynecologic cancer
* Hysterectomy not carried out using laparoscopy
* Fimbriated end missing or damaged or impossible for pathologist to analyze

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Female patients who underwent benign laparoscopic hysterectomy with systematic salpingectomy
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2014-01-31 (Actual); Primary Completion 2016-01-31 (Actual); Study Completion 2016-01-31 (Actual)

PRIMARY OUTCOMES:
Histopathologic tube anomalies | day 1 of surgery
  Prevalence of histopathologic tube anomalies (Serous Tubal Intraepithelial Carcinoma STIC or tumor protein 53 (p53) lesion)

CONTACTS AND LOCATIONS:
Overall Officials: Gautier Chene, PhD, Principal Investigator — Hospices Civils de Lyon (Hôpital Femme Mère Enfant)